CLINICAL TRIAL: NCT01606657
Title: Is Routine Irrigation of Cutaneous Abscesses Necessary?
Brief Title: Irrigation Versus no Irrigation for Cutaneous Abscess
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Brian Chinnock, Associate Clinical Professor of Emergency Medicine, Director of Coding/Reimbursement, University of California, San Francisco
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10012010
Record Dates: First submitted 2012-05-21; First posted 2012-05-28 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Cutaneous Abscess
Keywords: I&D; Abscess; Irrigation; Cutaneous Abscess
MeSH Terms: conditions — Abscess | interventions — Therapeutic Irrigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Irrigation (Active Comparator): THE PATIENT IS TO HAVE IRRIGATION OF THE ABSCESS WITH NORMAL SALINE AS PART OF THE I&D PROCEDURE
  Interventions: Procedure: Irrigation
- No Irrigation (Placebo Comparator): THE PATIENT IS NOT TO HAVE IRRIGATION OF THE ABSCESS AS PART OF THE I&D PROCEDURE
  Interventions: Other: No Irrigation

INTERVENTIONS:
Procedure: Irrigation — The patient will receive irrigation as a part of their wound care
  Arms: Irrigation
Other: No Irrigation — The patient will not receive irrigation as part of their wound care
  Arms: No Irrigation

SUMMARY:
In this study, the investigators are trying to find out if washing out the abscess (pocket of pus) with fluid will help, instead of only taking out the pus. Your care will be the same as usual, except that you will be selected randomly to have your abscess washed out with fluid, or not.

DETAILED DESCRIPTION:
Irrigation of the abscess cavity is commonly described as part of the procedure of incision and drainage of cutaneous abscesses (1-4). Despite this, there are no randomized controlled trials that demonstrate the benefit of irrigation in treatment of these abscesses. Potential disadvantages of irrigation include increased procedural time, pain, increased cost with sterile irrigation solutions and materials to capture the irrigation effluent, and increased risk of microbiologic contamination of the surrounding area. The goal of this study is to examine patients undergoing incision and drainage of cutaneous abscesses to determine if irrigation of the abscess cavity affects the need for further interventions.

ELIGIBILITY:
Inclusion Criteria:

1. All patients 18 years of age and above
2. Patients that require a cutaneous abscess incision and drainage

Exclusion Criteria:

1. Unable to return for 48-hour followup.
2. Patients being admitted to the hospital or going to the operating room for incision and drainage
3. Pregnant patients
4. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2010-08; Primary Completion 2014-09 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Patients needing further treatment after irrigation for I&D | 7 day phone follow-up
  Percentage of patients needing further treatment i. Further treatment defined as
  1. Repeat I&D
  2. Addition of an antibiotic (as new or to a pre-existing antibiotic)
  3. Admission to hospital for cutaneous abscess-related problem
     1. Abscess
     2. Cellulitis
     3. Septic arthritis
     4. Sepsis

SECONDARY OUTCOMES:
VAS is correlated with decreased pain after I&D | two years
  1) VAS post procedure pain score

CONTACTS AND LOCATIONS:
Overall Officials: Brian Chinnock, MD, Principal Investigator — UCSF, Community Regional Medical Center
Locations (1):
- Community Regional Trauma and Burn Center, Fresno, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Malley GF, Dominici P, Giraldo P, Aguilera E, Verma M, Lares C, Burger P, Williams E. Routine packing of simple cutaneous abscesses is painful and probably unnecessary. Acad Emerg Med. 2009 May;16(5):470-3. doi: 10.1111/j.1553-2712.2009.00409.x. Epub 2009 Apr 10. PMID 19388915
- [Background] Abraham N, Doudle M, Carson P. Open versus closed surgical treatment of abscesses: a controlled clinical trial. Aust N Z J Surg. 1997 Apr;67(4):173-6. doi: 10.1111/j.1445-2197.1997.tb01934.x. PMID 9137156
- [Background] Llera JL, Levy RC. Treatment of cutaneous abscess: a double-blind clinical study. Ann Emerg Med. 1985 Jan;14(1):15-9. doi: 10.1016/s0196-0644(85)80727-7. PMID 3880635
- [Background] Stewart MP, Laing MR, Krukowski ZH. Treatment of acute abscesses by incision, curettage and primary suture without antibiotics: a controlled clinical trial. Br J Surg. 1985 Jan;72(1):66-7. doi: 10.1002/bjs.1800720125. PMID 3881155